CLINICAL TRIAL: NCT01638182
Title: Comparison of Effects of Nutritional Doses Vitamin K1 and K2 on Carboxylation
Brief Title: Biocomparison Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-3-018
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Bone Health; Vascular Health
Keywords: phylloquinone,; menaquinone-7; vitamin K-status; efficacy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- vitamin K1 capsules (Active Comparator): 27 participants received for three months 1 vitamin K1-capsule per day containing 52 µg of K1
  Interventions: Dietary Supplement: Vitamin K1-capsules
- Vitamin K2-capsules (Active Comparator): 27 participants received for three months 1 vitamin K2-capsule per day containing 75 µg of MK-7.
  Interventions: Dietary Supplement: Vitamin K2-capsules
- Placebo capsules (Placebo Comparator): 27 participants received for 3 months 1 placebo capsule per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — 27 participants received for three months 1 placebo capsule per day
  Arms: Placebo capsules
Dietary Supplement: Vitamin K1-capsules — 27 participants received for 3 months 1 vitamin K1-capsule per day containing 52 µg of K1/day
  Arms: vitamin K1 capsules
Dietary Supplement: Vitamin K2-capsules — 27 participants received for 3 months 1 vitamin K2-capsule per day containing 75 µg of MK-7.
  Arms: Vitamin K2-capsules

SUMMARY:
The effects of two vitamin K-forms on carboxylation of the vitamin K-dependent proteins osteocalcin and matrix-gla protein will be compared after supplementing these vitamins in a nutritional dose range.

The investigators hypothesized that MK-7 is more effective than K1 at a dose comparable to the RDA of vitamin K.

DETAILED DESCRIPTION:
Vitamin K is a group name for the naturally occurring phylloquinone (K1) and menaquinones (MK-n; K2). The latter can be subdivided into the short-chain (e.g. MK-4) and the long-chain (e.g. MK-7, MK-8, and MK-9) menaquinones. Earlier studies have shown that high vitamin K intake leads to improved bone and vascular health by increased carboxylation of vitamin K-dependent proteins in these tissues. In the dietary range, MK-7 has been suggested to be the most effective cofactor for the carboxylation of Gla-proteins, such as osteocalcin (OC) and matrix-Gla protein (MGP).Until now, no randomized controlled trial has compared the efficacy of K1 versus MK-7 in a nutritional dose range. The investigators are therefore interested to compare the effects of K1 and MK-7 on OC and MGP carboxylation after supplementing these vitamins at a dose not exceeding the RDA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, aged between 20-80 years
* Normal body weight and height (18.5 kg/m2 < BMI < 30 kg/m2)
* Stable body weight (weight gain or loss < 3 kg in past 3 mo)
* Written consent to take part in the study
* Agreement to adhere to dietary restrictions required by the protocol

Exclusion Criteria:

* Abuse of drugs and/or alcohol
* Use of vitamin supplements containing vitamin K
* Pregnancy
* (a history of) metabolic or gastrointestinal diseases, e.g. hepatic or renal disorders, osteoporosis
* Chronic degenerative and/or inflammatory diseases, e.g. diabetes mellitus, cancer, cardiovascular disease
* Use of oral anticoagulants, drugs or hormones that influence bone metabolism
* Corticoid treatment
* Subjects with anaemia or subjects who recently donated blood or plasma
* Systemic treatment or topical treatment likely to interfere with coagulation metabolism (salicylates, antibiotics)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
carboxylation of osteocalcin | 12 weeks
  The primary objective of the study is to compare the effects of K1 and MK-7 on circulating ucOC levels after supplementing these vitamins at a nutritional dose.

SECONDARY OUTCOMES:
carboxylation of matrix-gla protein | 12 weeks
  The secondary objective of the study is to compare the effects of K1 and MK-7 on circulating ucMGP, which is emerging as a biomarker of arterial calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — VitaK BV Maastricht University
Locations (1):
- VitaK BV / Maastricht University Medicial Center, Maastricht, Netherlands